CLINICAL TRIAL: NCT03460262
Title: Negative Pressure Wound Therapy for Prevention of Groin Infection Following Vascular Surgery in High Risk Patient: a Randomized Control Study
Brief Title: Negative Pressure Wound Therapy for Prevention of Groin Infection Following Vascular Surgery
Acronym: PICO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/483
Record Dates: First submitted 2018-03-05; First posted 2018-03-09 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Infection Wound
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard dressing-Cutiplast® (Active Comparator)
  Interventions: Device: Standard cutiplast®
- Negative pressure wound therapy-PICO® (Experimental)
  Interventions: Device: PICO®

INTERVENTIONS:
Device: Standard cutiplast® — Our standard dressing consists in a usual ready-to-use Smith and Nephew Cutiplast®. This dressing is open 48 hours after the operation (CDC recommendation) for the first time and then changed every day after wound disinfection.
  Arms: Standard dressing-Cutiplast®
Device: PICO® — PICO® is a negative pressure wound therapy consisting in a 4 layers ready-to-use dressing connected to a small console, responsible for the aspiration. The system is canister free. The fluid drained from the wound is lost by evaporation for 80% of it and only 20% remains in the dressing. This permits to the dressing to be kept in place for maximum 7 days. The wound is not checked during the hospital stay, allowing the patient to leave the hospital earlier after the operation.
  Arms: Negative pressure wound therapy-PICO®

SUMMARY:
Surgical site infection in vascular surgery is a relatively common event with reported incidence as high as 43%. When considering the groin alone, the incidence is around 20% (30% when considering any wound complication). This complication may sometimes lead to heavier complication (leg amputation, longer hospital stay, high costs…) and affects the early postoperative quality of life of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Every high-risk patient (meeting one of the criteria of table I) undergoing vascular surgery with groin incision (without ongoing infection)

Exclusion Criteria:

* Patients who need a transverse incision before EndoVascular Aortic Repair procedure, considering that in our experience surgical site infection almost never occurs after these procedures and patients with mental incapacities.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2018-03-15 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-11-30 (Estimated)

PRIMARY OUTCOMES:
The rate of wound complications | at one year

CONTACTS AND LOCATIONS:
Overall Officials: Parla Astarci, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques Universitaires Saint-Luc, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
It is not decided yet.

REFERENCES:
- [Derived] Correia RM, Nakano LC, Vasconcelos V, Cristino MA, Flumignan RL. Prevention of infection in peripheral arterial reconstruction of the lower limb. Cochrane Database Syst Rev. 2025 Oct 29;10(10):CD015022. doi: 10.1002/14651858.CD015022.pub2. PMID 41159585